CLINICAL TRIAL: NCT05327582
Title: A Phase I/II, Open-label, One-arm, Single-center Study to Evaluate the Safety and Efficacy of the PLENA Regimen in Subjects With Unresectable Pancreatic Cancer or Biliary Tract Cancer
Brief Title: An Open-label, Phase I/II Study of PLENA Regimen in Patients With Unresectable Pancreatic Cancer or BTC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Principal Investigator, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-070
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Pancreatic Cancer; Biliary Tract Cancer
Keywords: unresectable; anti-PD-L1 antibody; lenvatinib; nab-paclitaxel
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms | interventions — durvalumab; lenvatinib; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLENA regimen (Experimental): Subject received PLENA regimen every 3 weeks until achieving a second assessable complete response or up to a maximum of 8 cycles. Treatment continued until progressive disease or intolerable toxicity, or withdrawal of consent.
  Interventions: Drug: Durvalumab; Drug: Lenvatinib; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Durvalumab — Administered intravenously, 1000 mg on day 1 in a 3-week cycle
Drug: Lenvatinib — Administered orally, 8mg/d once daily in a 3-week cycle
Drug: Nab paclitaxel — Administered intravenously, 180-220 mg/m2 on day1 in a 3-week cycle

SUMMARY:
Immunotherapy of cancer based on PD-1/PD-L1 blockade has prompted a revolution in cancer clinical management, albeit as yet immunotherapy-based treatment approaches in pancreatic cancer and biliary tract cancer (BTC) remain to have proven value, highlights the urgency for designing novel therapeutic strategies to combat these deadly diseases. The immunomodulatory effect of lenvatinib (Lenvatinib is an oral multi-kinase inhibitor) on tumor microenvironments may contribute to antitumor activity of immune checkpoint blockade. This one-arm, phase I/II study is designed to assess the safety and efficacy of the combined regimen of Durvalumab (anti-PD-L1 antibody), Lenvatinib and Paclitaxel albumin (nab-paclitaxel).

ELIGIBILITY:
Inclusion Criteria:

1.Subjects must have histologically proven unresectable pancreatic cancer or biliary tract cancer 2.18 to 75 years old. 3.Life expectancy of at least 6 months. 4.Eastern Cooperative Oncology Group performance status 0-2. 5.Subjects must have at least one measurable lesion ≥ 1 cm as defined by response criteria.

6.Subjects with Anti-PD-1/L1 antibody treatment history are eligible which must be disease progression.

7.Adequate organ function. 8.Participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drug.

Exclusion Criteria:

1. Subjects with any autoimmune disease or history of syndrome that requires corticosteroids or immunosuppressive medications.
2. Serious uncontrolled medical disorders or active infections, pulmonary infection especially.
3. Prior organ allograft.
4. Women who are pregnant or breastfeeding.
5. Women with a positive pregnancy test on enrollment or prior to investigational product administration.
6. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-04-12 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with treatment-related adverse events (AEs) | 6 months
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0. AEs were considered to be treatment-related if they had started or worsened within the interval from first study drug administration until the follow-up visit.
Object response rate (ORR) | 12 months
  ORR is defined as the proportion of subjects who achieved a partial response (PR) or complete response (CR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 12 months
  DCR is defined as the proportion of subjects who achieved a stable disease (SD), partial response (PR) or complete response (CR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Progression-free survival (PFS) | 12 months
  PFS time was measured from study entry to the first documentation of disease progression or death. Disease progression was determined per the RECIST V1.1.
Overall survival (OS) | 24 months
  OS time was measured from the study entry to the date of death.
Number of participants with laboratory test abnormalities | 12 months
  The laboratory tests of serum cytokines and chemokines will be performed on day 1 of each cycle, and the abnormality will be determined by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, Dr, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided